CLINICAL TRIAL: NCT07245407
Title: A Multi-center Longitudinal Observation Translational Study to Evaluate Phenotypes, Endotypes and Biomarkers in Chinese Patients With NCFBE
Brief Title: A Translational Study for Phenotyping and Endotyping Chinese Patients With NCFBE
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9186R00001
Record Dates: First submitted 2025-09-29; First posted 2025-11-24 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Non-cystic Fibrosis Bronchiectasis
Keywords: NCFBE

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy control cohort: Healthy controls will include at least 20 healthy participants aged 30 years or older, with no clinically significant lung disease or chronic lung disease.
  Interventions: Other: Participant Follow-up
- Bronchiectasis cohort: A total of up to 300 NCFBE patients (males and females aged 18 years or older) will be recruited and enrolled into the study. Patient numbers are mainly based on feasible situation.
  Approximately 30% of NCFBE patients in the study will be required to have had at least 2 exacerbations in the past 12 months.
  Interventions: Other: Participant Follow-up

INTERVENTIONS:
Other: Participant Follow-up — This is a longitudinal multi-center, observational, translational study which includes patients with a physician diagnosis of NCFBE by chest HRCT and healthy controls (at baseline only).
  This study will consist of a baseline visit, a 6-month (site visit or telephone visit) and a 12-month visit as well as planned unscheduled visits for exacerbation events and one optional visit for bronchoscopy.Healthy participants will be only enrolled in the baseline visit and bronchoscopy visit.

SUMMARY:
Background/Rationale:

Non-cystic fibrosis bronchiectasis (NCFBE) is a chronic respiratory disease characterized by a clinical syndrome of chronic productive cough and recurrent respiratory infections in the presence of abnormal and permanent dilation of the bronchi. Recent epidemiological studies have clearly shown that the prevalence and incidence of NCFBE are quickly rising both in high- and low-income countries. With the increase of prevalence, bronchiectasis brings huge medical and economic burden to the society.

Recently published Chinese Bronchiectasis Registry study (BE-China) data showed that Chinese bronchiectasis patients exhibit unique clinical characteristics when compared to western countries. The proportion of post-infective causes and tuberculosis in China was twice that of the European Multicenter Bronchiectasis Audit and Research Collaboration (EMBARC) cohort. Moreover, Chinese patients had a lower FEV1% of predicted value, and a higher proportion of obstruction compared to the EMBARC cohort. Pseudomonas aeruginosa (PsA) was the most common pathogen in both cohorts. Chinese patients exhibited a higher frequency of hospitalization compared to the EMBARC cohort (57.2% vs 26.4%); however, unlike the frequency of hospitalization, Chinese patients had fewer exacerbations in the year before enrollment compared to the EMBARC cohort, with most having only one exacerbation. The proportion of patients with three or more exacerbations was much higher in the EMBARC cohort than in China (12.3% vs 38.8%). Except for Aspergillus fumigatus, the positive culture rates of other pathogens were much higher in the EMBARC cohort than in China.

Significant difference in aetiology and clinical phenotypes of NCFBE has been demonstrated by many registry studies conducted in different geographical regions including EMBARC and BE-China. However, the biological processes and mechanisms driving the disease development, so-called "endotypes", have not been fully investigated within the patient populations in these studies. It is remaining unknown that if these differences reported in clinical phenotypes were truly caused by or linked to different endotypes in NCFBE.

In this study, the investigator will perform biomarker assessments and multi-omics analysis on NCFBE patients and healthy participants in China to validate the link of disease pathways to pathophysiological features and uncover the molecular endotypes behind clinical phenotypesof Chinese patients with NCFBE.

ELIGIBILITY:
Inclusion Criteria:

Healthy control cohort:

· Age ≥30 years

Bronchiectasis cohort:

* Capable of giving signed informed consent.
* Participant must be ≥18 years of age, at the time of signing the ICF.
* Able to perform acceptable lung function testing according to ATS/ERS 2019 acceptability criteria.
* Able and willing to comply with the requirements of the protocol including ability to read, write, be fluent in the translated language of all participants facing questionnaires used at center, and use electronic devices (e.g. FENO and spirometry).
* Documented physician-diagnosed bronchiectasis: with a clinical history consistent with bronchiectasis (chronic cough and daily sputum production etc.) and having performed chest HRCT indicating bronchiectasis.
* Remaining clinically stable upon recruitment. Patients with exacerbations are allowed to be enrolled into the registry at least 4 weeks after antibiotic discontinuation.

Exclusion Criteria:

Healthy control cohort:

* Any respiratory diagnosis (asthma, COPD, bronchiectasis, pulmonary fibrosis or any other chronic respiratory condition requiring regular treatment).
* Inflammatory conditions including rheumatoid arthritis, inflammatory bowel disease, any other connective tissue disease.
* Active malignancy excluding non-melanoma skin cancer.
* Antibiotic treatment for an acute respiratory tract infection in the previous 4 weeks or current sinusitis.
* Any contraindication to study procedures including bronchoscopy.
* Current smoking or smoking in the preceding 3 months.
* Treatment with anti-coagulants.

Bronchiectasis cohort:

* Traction bronchiectasis associated with interstitial lung disease or other pulmonary disorders (e.g., pulmonary fibrosis and cystic fibrosis).
* Primary diagnosis of another pulmonary condition, including COPD, asthma. Patients with a secondary diagnosis of these pulmonary diseases will be allowed to participate as long as bronchiectasis is considered by the investigator to be the primary diagnosis.
* Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematological, psychiatric, or major physical impairment that is not stable in the opinion of the investigator and could:
* Affect the safety of the participant throughout the study
* Influence the findings of the study or the interpretation
* Impede the participant's ability to complete the entire duration of study
* The participant has a history of alcohol or drug abuse within the past year, which, in the opinion of the responsible physician, contra-indicates their participation.
* Active malignancy excluding non-melanoma skin cancer.
* Participants is female who is pregnant or lactating or up to 6 weeks post-partum or 6 weeks cessation of breastfeeding.
* The participant has an altered mental status at the time of informed consent.
* History or current evidence of an upper or lower respiratory infection or symptoms(including common cold) within 2 weeks of baseline assessments
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study center).
* Terminal disease and/or organ failure or participants otherwise considered not appropriate for the study participation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy controls will include at least 20 healthy participants aged 30 years or older, with no clinically significant lung disease or chronic lung disease.
  A total of up to 300 NCFBE patients (males and females aged 18 years or older) will be recruited and enrolled into the study. Patient numbers are mainly based on feasible situation.
  Approximately 30% of NCFBE patients in the study will be required to have had at least 2 exacerbations in the past 12 months.
  A subset of 60 NCFBE patients and 20 healthy participants is planned for an optional bronchoscopy assessment.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2027-07-29 (Estimated); Study Completion 2027-07-29 (Estimated)

PRIMARY OUTCOMES:
FEV1/FVC% | 12 month
  Evaluation of lung function
FEF25-75 L/s | 12 month
  Evaluation of small airway function
FENO ppb | 12 month
  Evaluation of airway inflammation: FENO.
HRCT | 12 month
  Evaluation of lung structure profile and change through radiological parameters.
cell percentage (%) | 12 month
  Measurement of immune cell (including but not limited to neutrophils and eosinophils) percentages in samples such as blood, sputum, and BALF.
Gene expression read counts by RNAseq | 12 month
  Functional and transcriptional characterization of airway immune cells, bronchial epithelial cells andsmooth muscle cells (optional).
Molecular deliverables | 12 month
  8-OHdG (8-Hydroxyguanosine) in different sample matrix including but not limited to serum, urine and sputum (ng/ml)
on-set age(years-old) | 12 month
  Risk factor assessment: on-set age(years-old)
Sex(M/F) | 12 month
  Risk factor assessment: Sex(M/F)
body mass index(kg/m^2) | 12 month
  Risk factor assessment: body mass index(kg/m^2)
comorbidities | 12 month
  Risk factor assessment: comorbidities
medical history | 12 month
  Risk factor assessment: medical history, especially TB history
smoking status(never/current/former) | 12 month
  Risk factor assessment: smoking status(never/current/former)
smoking pack years(pack/year) | 12 month
  Risk factor assessment: smoking pack years(pack/year)
Sputum microbiology (CFU) | 12 month
  Bronchiectasis aetiology evaluation
Historical Exacerbation | 12 month
  Risk factor assessment: exacerbation number in the previous year
BSI score | 12 month
  Evaluation of ronchiectasis disease severity: BSI score(0-4 mild,5-8 moderate, ≥9 severe)
QoL-B-RSS | 12 month
  Evaluation of quality of life: Patient reported outcome: QoL-B-RSS (0-100, higher score stands for lower symptom burden and higher quality of life)
BHQ | 12 month
  Evaluation of quality of life: Patient reported outcome: BHQ(10-70,higher score stands for higher symptom burden and pooer quality of life )
BEST | 12 month
  eDiary: BEST(MCID 4 points may standfor an exacerbation.)
Treatment pattern | 12 month
  Evaluation of treatment pattern: inhaled antibiotic, macrolide, and mucoactive drugs,etc.
Exacerbation assessment | 12 month
  Exacerbation assessment: number of exacerbations per patient per year
Cell counts (10^9/L) | 12 month
  Measurement of immune cell (including but not limited to neutrophils and eosinophils) counts in samples such as blood, sputum, and BALF.
Exacerbation assessment | 12 month
  Exacerbation assessment: number of exacerbations lead to hospitalization per patient per year

CONTACTS AND LOCATIONS:
Locations (1):
- Huadong Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org